CLINICAL TRIAL: NCT07251673
Title: Longitudinal Study of Phenotypic and Developmental Severity in Patients With Dravet Syndrome With SCN1A Gene Mutation
Acronym: LONG-DS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Encoded Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP241685; 2024-A02640-47 (Other: ANSM)
Record Dates: First submitted 2025-08-19; First posted 2025-11-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Dravet Syndrome
Keywords: Dravet syndrom; epilepsy
MeSH Terms: conditions — Epilepsies, Myoclonic; Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — An extra tube of blood taken during a blood test for metabolomics for metabolomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dravet syndrom Cohort: Blood sample for metabolomic analysis and scale

SUMMARY:
Dravet syndrome with SCN1A gene mutation is a developmental and epileptic encephalopathy characterized by treatment-resistant epilepsy and global developmental delay.

Despite the considerable attention recently Dravet syndrome (DS) in drug development, studies characterising the progression of the neurodevelopmental phenotype over time remain limited. In particular, many previous studies of natural history studies have been of short duration or have focused only on a subgroup of the paediatric population.

This prospective natural history study is being conducted to define more precisely the neurodevelopmental trajectory of SCN1A-positive Dravet syndrome in patients aged aged 6 months to 21 years with SCN1A mutations. The study will examine these characteristics over a 4-year period using standardised assessments. The study will also explore potential metabolomic biomarkers and their relationship with clinical outcomes.

DETAILED DESCRIPTION:
A prospective cohort to document the evolutionary trajectory over a 4-year period of patients with Dravet syndrome with a confirmed pathogenic or probably pathogenic variant in the SCN1A gene aged between 6 months and 21 years.

Pre-selection/eligibility stage Patients and their legal representatives will be contacted by an investigator. Inclusion and non-inclusion criteria will be assessed to confirm the participant's eligibility, allowing entry into the study and completion of the baseline assessment. Following a discussion of the objectives, risks and benefits of the study, the patient's non-objection to taking part in the research will be obtained, together with the patient's assent, if applicable.

Baseline assessment (Year 0)

An initial visit will be organized to collect demographic, historical and clinical data, and to carry out :

1. A detailed medical assessment (age, sex, history of seizures genetic diagnosis, co-morbidities, current treatments).
2. The Vineland-3 (parental module), analyzed by a psychologist
3. GMFM-66 for motor functions (by a physiotherapist).
4. CGI-S scale (clinician and carer)
5. An additional tube of blood taken during a blood test for metabolomics analysis (including serum GABA).
6. Bayley-IV (up to 8 years, depending on chronological or developmental age).

Annual visits (Years 1 to 4)

Annual assessments will be carried out to document clinical progress and will include:

1. A medical update (new diagnoses, types and frequency of seizures, treatments).
2. The same assessment tools as at the initial visit (Vineland-3, GMFM-66, CGI-S, Bayley-IV).
3. The CGI-I scale to measure changes since the previous visit.
4. An extra tube of blood taken during a blood test for metabolomics for metabolomic analysis.
5. The collection of data from medical examinations carried out as part of the treatment.

End of the study After four annual visits following the baseline assessment, the participant will complete the study. A final report will be drawn up to document the clinical and functional evolution of Dravet syndrome over a 4-year period

ELIGIBILITY:
Inclusion Criteria:

* The patient or his/her legal representative must be able to give informed consent for participation in the study.
* The participant or legal representative are able (in the opinion of the investigator) to comply with the research protocol.
* Patient (male/female) between 6 months and 21 years of age inclusive at the time of consent.
* The patient has a confirmed pathogenic or probably pathogenic variant of the SCN1A gene demonstrated by a genetic test.
* The patient had normal development prior to the onset of the first seizure.
* The patient had an onset of epileptic seizures between the ages of 3 and 15 months inclusive.
* The patient is receiving at least one of the following anti-epileptic drugs prior to consent: brivaracetam, clobazam, cannabidiol, fenfluramine, levetiracetam, sodium valproate, stiripentol, topiramate

Exclusion Criteria:

* The patient has a copy number variation of the SCN1A gene affecting other genes, including a microdeletion of SCN1A.
* The patient has a mutation in the SCN1A gene on both alleles.
* The patient has a known or clinically suspected pathogenic mutation in a gene associated with epilepsy other than the SCN1A gene.
* The patient has a concomitant genetic mutation or clinical comorbidity deemed likely to disrupt the typical phenotype of Dravet syndrome.
* The patient has a known gain-of-function mutation, defined by functional studies, including p.Thr226Met.
* The patient has a history of neurodevelopmental abnormality prior to the onset of seizures, based on the medical record.
* The patient has been seizure free for a period of one year prior to informed consent.
* The patient has, at any time, taken antiepileptic drugs with a worsening effect for 6 consecutive weeks or more, including: carbamazepine, eslicarbazepine, lacosamide, lamotrigine, oxcarbazepine, phenytoin (chronic oral administration), tiagabine and vigabatrin.
* The patient has already received innovative therapies such as antisense ologonucleotides, gene therapy or cell therapy.
* The patient has a structural abnormality on brain imaging (MRI or CT scan) which the principal investigator considers to be an epileptogenic lesion.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 6 months to 21 years with Dravet syndrome due to a pathogenic or probably pathogenic variant of the SCN1A
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Score of scale Vineland-3 | Up to 4 years
  Change in adaptive function measured by the Vineland-3 over time at 1, 2, 3 and 4 years follow-up (160 is the maximum score and 20 is the minimum score - the higher score is the better outcome)

SECONDARY OUTCOMES:
Score of scale Gross Motor Function Measure-66 (GMFM-66) | Up to 4 years
  Changes in motor function and activity measured by the GMFM-66 Max value:201 Min value:0 Higher score is the better outcome
Score of scale Bayley-IV sub-domains | Up to 4 years
  To study the evolution of adaptive capacities over time in Dravet syndrome by changes in raw score for Bayley-IV sub-domains (160 is the maximum score and higher score and 40 is the minimum score - the higher score is the better outcome)
Average Clinical Global Impressions (CGI) scale score at each age | Up to 4 years
  To understand the severity of Dravet syndrome with SCN1A mutation (Rating by the investigator, where 1 is the best outcome and 7 is the worst outcome)
Score of improvement scale | Up to 4 years
  To understand the severity of Dravet syndrome with SCN1A mutation and how this severity changes with age. (Rating by the investigator, where 1 is the best outcome and 7 is the worst outcome)
Dosage of serum GABA | Up to 4 years
  Average serum GABA level in each age group

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Auvin, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, Ap-hp / DRCI, France